CLINICAL TRIAL: NCT05402657
Title: The Randomised Controlled Trial of Frontoparietal and Temporoparietal Electroconvulsive Therapy (ECT) for Severe Depression: The RAFT ECT Study
Brief Title: The RAFT ECT Study
Acronym: RAFT-ECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Ramsay Clinic Albert Road, Australia (Unknown); Ramsay Clinic Lakeside, Australia (Unknown); Ramsay Clinic Northside, Australia (Unknown); Gold Coast Hospital and Health Service (Other Government); Augusta University (Other); Medical University of South Carolina (Other); The University of New South Wales (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X22-0018; APP1159769 (Other Grant/Funding Number: NHMRC); RG180233 (Other: UNSW project number)
Record Dates: First submitted 2022-05-05; First posted 2022-06-02 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Episode
Keywords: Severe depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Memory; Electroconvulsive therapy; Randomised clinical trial
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors completing assessments of mood (primary outcome) will be blinded to the participant's treatment allocation until the database is locked and the primary analysis completed. Hospital ward personnel, if not involved in the delivery of ECT, will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frontoparietal ECT Group (Experimental): Participants will receive ultrabrief right unilateral ECT with a frontoparietal placement of ECT electrodes.
  Interventions: Procedure: Frontoparietal Ultrabrief Right Unilateral (UBRUL-FP) electroconvulsive therapy
- Temporoparietal ECT Group (Active Comparator): Participants will receive ultrabrief right unilateral ECT with the conventional temporoparietal placement of ECT electrodes.
  Interventions: Procedure: Temporoparietal Ultrabrief Right Unilateral (UBRUL-TP) electroconvulsive therapy

INTERVENTIONS:
Procedure: Frontoparietal Ultrabrief Right Unilateral (UBRUL-FP) electroconvulsive therapy — UBRUL-FP involves ultrabrief right unilateral ECT delivered using a novel frontoparietal montage, where the anterior electrode is shifted frontally to a position above the midpoint of the right eye to avoid temporal lobe stimulation (and reduce memory side effects). UBRUL-FP will be delivered using standard ECT devices.
  Arms: Frontoparietal ECT Group
Procedure: Temporoparietal Ultrabrief Right Unilateral (UBRUL-TP) electroconvulsive therapy — UBRUL-TP is the standard form of ultrabrief right unilateral ECT, using the conventional temporoparietal (d'Elia) electrode placement, where the anterior electrode is placed over the right temporal lobe. UBRUL-TP will be delivered using standard ECT devices.
  Arms: Temporoparietal ECT Group

SUMMARY:
Severe depression is devastating for those affected and is often associated with significant risk of suicide. Electroconvulsive therapy (ECT) is a highly effective acute treatment for severe depression, but its use and acceptability are limited by cognitive side effects. Of these, retrograde memory loss is most concerning, and can be long-term. The introduction of ultrabrief right unilateral (UBRUL) ECT into clinical practice has been an important step in reducing the risk of memory impairment, but significant deficits still occur.

A new form of UBRUL ECT which utilises a Frontoparietal electrode placement represents a further development. Preliminary data suggest that Frontoparietal UBRUL has good efficacy and less cognitive side effects than UBRUL given using the conventional Temporoparietal electrode placement. Designed as a pivotal trial, this protocol will be the first RCT comparing these two forms of ECT, producing the rigorous efficacy and safety data required to change clinical practice/policy.

This is a multicentre, parallel group RCT with 1:1 allocation ratio between Frontoparietal (intervention) and Temporoparietal (comparator) forms of UBRUL ECT. Participation will involve receiving randomised acute ECT under blinded conditions during the randomised acute treatment period (typically around 4 weeks), then completion of a 24-week follow-up period which commences after the cessation of all acute ECT. The study protocol aims to provide 12 randomised acute ECT treatments, though the number of treatments (and hence the length of the randomised acute treatment period) can be adjusted by the participant's own treating/admitting psychiatrist according to their clinical judgement.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis* of major depressive episode (unipolar or bipolar)
* HRSD-17 score ≥ 17 at Screening
* At least 18 years old
* Able to tolerate washout of prohibited medications and restriction on benzodiazepine dosage, as determined by patient's own treating psychiatrist.
* ECT indicated for treatment of depression, as determined by own treating referring psychiatrist and confirmed by research evaluations (e.g., diagnosis of depression)
* Willing and able to participate in research and comply with study requirements
* Sufficient proficiency in spoken English to ensure validity of neuropsychological testing (e.g., worked or studied in an English-speaking context or equivalent)

Exclusion Criteria:

* History of schizophrenia, schizoaffective disorder, other [non-mood disorder] psychosis, or rapid cycling bipolar disorder (DSM-5 diagnoses*)
* Current manic episode, hypomanic episode, or major depressive episode with mixed features (DSM-5 diagnoses*)
* Alcohol or substance use disorder (other than caffeine or nicotine) present in the past month, or is likely to be present during the 24-week study period as determined by study physician evaluation
* Diagnosis of amnestic disorder, dementia, delirium, or epilepsy, as determined by study physician evaluation and medical history
* Central nervous system disease or brain injury that has resulted in significant cognitive impact, as determined by study physician evaluation and medical history
* Serious or unstable medical condition, as determined by study physician evaluation and medical history
* If female of childbearing potential: a) pregnancy as determined by pregnancy urine screen
* Completed an acute course of ECT during the past 2 months, as determined by treatment history
* Received any ECT during the past 2 weeks
* Failed an adequate course of ECT (i.e., 8 ECT treatments ) in the current depressive episode
* Patients who are prisoners, and those who lack capacity to make medical decisions (as judged by their own treating psychiatrist)
* Currently enrolled in another interventional clinical trial
* Currently using another investigational device or product

  * DSM-5 psychiatric diagnoses will be assessed and confirmed using the Mini International Neuropsychiatric Interview (MINI; Sheehan et al., 1998) Version 7.0.2 for DSM-5, administered by research team members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms as Assessed by Hamilton Rating Scale for Depression-17 | From baseline to end of randomized acute treatment (typically 4 weeks)
  The Hamilton Rating Scale for Depression-17 has a range of 0-52. Lower scores represent mild depression to no depression at all.

SECONDARY OUTCOMES:
Change in Depressive Symptoms as Assessed by Hamilton Rating Scale for Depression-17 | From end of acute ECT treatment up to 24-week follow-up
  The Hamilton Rating Scale for Depression-17 has a range of 0-52. Lower scores represent mild depression to no depression at all.
Autobiographical Memory Interview-Short Form (AMI-SF) Consistency Scores | From Baseline to end of randomized acute treatment (typically 4 weeks)
  In the Autobiographical Memory Interview-Short Form, participants are graded on the consistency of their answers between baseline and subsequent time-points. The maximum consistency score is 100 percent, with lower percentages representing increasing inconsistency in retrospective autobiographical memory function.
Clinical Global Impression-Severity (CGI-S) | From baseline to end of randomized acute treatment (typically 4 weeks)
  The Clinical Global Impression-Severity measure is a 7-point scale where a clinician rates the severity of a patient's illness in comparison to the clinician's experience with patients who have the same diagnosis. The ratings range from 1 indicating normal, not at all ill to 7 suggesting they are among the most extremely ill patients.
Clinical Global Impression-Improvement (CGI-I) | Through the randomized acute ECT treatment period (typically 4 weeks)
  The Clinical Global Impression-Improvement is a measure where a clinician assesses how much the patient's illness has improved or worsened in comparison to baseline. The "improved" version being used in this trial (Kadouri, Corruble & Falissard, 2007) is a 13-point scale with ratings which range from 6 ('ideal improvement') to -6 (maximum deterioration).
Suicidality score | From baseline to end of randomized acute treatment (typically 4 weeks)
  Assessed by examining scores on item 3 (suicidality) of the Hamilton Rating Scale for Depression (which range from 0 to 4, where higher scores indicate more severe and/or persistent suicidality) and scores on the suicidal ideation subscale of the Columbia
Post ECT reorientation time | After ECT sessions 3 and 6, which typically occur at the end of week 1 and week 2 in the randomised acute treatment phase.
  Post ECT reorientation time is the time taken to recover orientation immediately after ECT in randomised treatment phase.
Change in mean neuropsychological function | From baseline to end of randomized acute treatment (typically 4 weeks)
  Assessed by a cognitive test battery.
Mental Health Questionnaire-14 (MHQ-14) | From baseline to end of randomized acute treatment (typically 4 weeks)
  The Mental Health Questionnaire-14 is a self-report quality of life instrument consisting of the mental health component of the Medical Outcomes Study questionnaire. This patient self-report measure contains 14 items in total, addressing symptoms of fatigue, anxiety and depression, and the impact of these symptoms on functioning. Scores on this measure range from 0 to 100, where higher scores indicate better quality of life.
Number of responders | From baseline to End of Randomized Acute Treatment (typically 4 weeks)
  Response is defined as a 50 percent reduction in depression severity from baseline, assessed using the Hamilton Rating Scale for Depression-17
Number of remitters | From baseline to end of randomized acute treatment (typically 4 weeks)
  Remission is defined as a score of ≤ 7 on the Hamilton Rating Scale for Depression-17.
Number of participants switched from randomized treatment to another form of acute ECT | After at least 8 randomized ECT treatments (typically after 3 weeks).
  Number of participants switched from randomized treatment to another form of acute ECT after receiving at least 8 randomized ECT.
Number of randomized ECT treatments given over the Acute Study Treatment Phase (RCT) | From baseline to End of Randomized Acute Treatment (typically 4 weeks)
  Number of randomized acute ECT treatments received by participants during the Acute Study Treatment Phase (RCT), compared between the groups.
Occurrence of adverse events and serious adverse events | From baseline and up to 24-week follow-up
  Occurrence of adverse events (AEs) and serious adverse events (SAEs) compared between the groups, based on treating them as binary outcomes (no/yes, e.g., whether participants experienced any given side effect/adverse event at least once) and as count outcomes (number of occurrences).

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, Principal Investigator — University of New South Wales; Anthony Rodgers, Study Director — The George Institute
Locations (7):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta University, Augusta, Georgia
  - Medical University of South Carolina, Charleston, South Carolina
- Australia (4):
  - Ramsay Clinic Northside, Sydney, New South Wales
  - Ramsay Clinic Lakeside, Warners Bay, New South Wales
  - Gold Coast University Hospital (GCUH), Gold Coast, Queensland
  - Ramsay Clinic Albert Road, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon request to the data custodian, subject to approval from the Trial Steering Committee and signing of data transfer agreements.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Loo C, Barreiros AR, Martin D, Dong V, George MS, McCall WV, Sarma S, Hopwood M, Weiss A, Bull M, Tuneu CM, Alonzo A, Hadzi-Pavlovic D, Rodgers A, Sahlem GL, Harvey AJ, Haldane K, Brettell L, Fitzgerald PB, Dokos S, Sackeim H. A Randomized Controlled Trial of Ultrabrief Right Unilateral ECT With Frontoparietal Versus Temporoparietal Electrode Placement for Severe Depression-The RAFT ECT Trial. J ECT. 2024 Dec 1;40(4):229-231. doi: 10.1097/YCT.0000000000001018. Epub 2024 Jul 5. No abstract available. PMID 38968425